CLINICAL TRIAL: NCT02285205
Title: A 24 Week, Multicenter, Prospective, Open-labeled, Single-arm, Exploratory Phase 4 Clinical Trial to Evaluate the Safety and Efficacy of Lobeglitazone in Decreasing Intrahepatic Fat Contents in Type 2 Diabetes With NAFLD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2014-0778
Record Dates: First submitted 2014-11-04; First posted 2014-11-06 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes; Non-alcoholic Fatty Liver Disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lobeglitazone (Experimental)
  Interventions: Drug: Oral administration of Lobeglitazone

INTERVENTIONS:
Drug: Oral administration of Lobeglitazone — Lobeglitazone 0.5mg/tablet, orally, 1 tablet once daily for 24 weeks

SUMMARY:
Lobeglitazone is highly selective peroxisome proliferator-activated receptor-gamma agonist that decreases insulin resistance in the periphery and liver resulting in increased insulin-dependent glucose disposal and decreased hepatic glucose output. In vivo, It demonstrates that Lobeglitazone improves even more glycemic and lipid control in comparison to rosiglitazone and pioglitazone. Currently, thiazolidinediones such as pioglitazone is the only drug which is considered as an effective therapeutic agent for improving non-alcoholic fatty liver disease (NALFD) in type 2 diabetes (T2D).

The aim of this multicenter, prospective, open-labeled, single-arm, exploratory phase 4 study is to evaluate the efficacy and safety of Lobeglitazone once daily for 24 weeks on intrahepatic fat contents assessed by transient elastography (fibroscan) in T2D with NAFLD.

Fifty subjects with T2D and NAFLD will take Lobeglitazone (0.5mg/tablet, orally, 1 tablet once daily) for 24 weeks.

Primary endpoint is changes from baseline in controlled attenuation parameters (CAP) measured by transient elastography (fibroscan) after treatment with Lobeglitazone.

Secondary endpoints are changes from baseline in glycemic profiles (HbA1c, Glycated albumin), Lipid parameters (Total Cholesterol, Triglycerides, HDL-C, LDL-C), Liver function parameters (AST, ALT, r-GT), and adverse events during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Type Ⅱ diabetes mellitus
2. Non-alcoholic fatty liver disease: subjects who have CAP(Controlled Attenuation Parameter) ≥ 250dB/m measured by transient elastography (fibroscan) at screening test
3. Age ≥ 20 years
4. Patients who have not been taking any oral hypoglycemic agent for more than 12 weeks with HbA1c 7.0 to 8.5% at screening test or who have been taking metformin monotherapy for at least 8 weeks with HbA1c 7 to 9% at screening test
5. Agreement with written informed consent

Exclusion Criteria:

1. Patients whose alcohol consumption >210g/week for males and 140g/week for females
2. chronic B viral hepatitis, chronic C viral hepatitis, Type I diabetes, or secondary diabetes
3. having a history of acute or chronic metabolic acidosis including diabetic ketoacidosis
4. patients who have been taking other oral hypoglycemic agents except metformin or insulin within recent 8 weeks
5. who experienced hypersensitivity reaction against metformin or glitazone drugs
6. who has been treated with corticosteroids for at least 14 days within 2 month prior to Screening
7. having a history of lactic acidosis
8. having genetic predispositions such as galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption
9. who are in condition of malnutrition, starvation, cachexia, severe infection, major trauma, hypopituitarism, or adrenal insufficiency
10. diagnosed with cancer within 2 years or having chemo or radiotherapy for cancer treatment
11. a history of drug abuse or chronic alcoholism
12. a history of heart failure (NYHA class III and IV) or uncontrolled arrhythmia
13. a history of acute cardiovascular or cerebrovascular disease within 12 weeks prior to Screening (unstable angina, myocardial infarction, transient ischemic attack, cerebral infarct, cerebral hemorrhage, coronary bypass, percutaneous coronary intervention)
14. Renal dysfunction: Serum creatinine greater than 1.5mg/dl for males and 1.4mg/dl for females.
15. Anemia less than 10.5g/dl for any reason
16. Pregnant women or nursing mothers
17. Fertile women who not practice contraception with appropriate methods
18. in treatment concomitant drug from other clinical trials within 4 weeks from enrollment
19. who did not agree with written informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
changes from baseline in controlled attenuation parameters (CAP) | 24 weeks
  Changes from baseline in controlled attenuation parameters (CAP) measured by transient elastography (fibroscan) after treatment with Lobeglitazone

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Department of Internal Medicine, Yonsei University College of Medicine, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Lee YH, Kim JH, Kim SR, Jin HY, Rhee EJ, Cho YM, Lee BW. Lobeglitazone, a Novel Thiazolidinedione, Improves Non-Alcoholic Fatty Liver Disease in Type 2 Diabetes: Its Efficacy and Predictive Factors Related to Responsiveness. J Korean Med Sci. 2017 Jan;32(1):60-69. doi: 10.3346/jkms.2017.32.1.60. PMID 27914133